CLINICAL TRIAL: NCT03187145
Title: A Cohort Study of Ultrasound Evaluation of Gastric Emptying in Diabetic Patients: a Comparison With Healthy Controls
Brief Title: Ultrasound Evaluation of Gastric Emptying in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: wch-160023
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic patients
- healthy control

SUMMARY:
This is a prospective cohort study. The main objective is to compare the frequency of a "full stomach" in the diabetic population compared to healthy controls 2 h after clear liquid and 6h after a light meal, and evaluate the mean gastric emptying time of clear liquid and light meal in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic and non-diabetic Patients scheduled for elective surgery aged 18 to 85years American Society of Anesthesia physical status classification I to III Body mass index < 40 kg/ cm2.

Exclusion Criteria:

* Pregnancy (currently or within the past 3 months) Previous surgery of the upper gastrointestinal tract Achalasia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be diabetic and non-diabetic patients whom are scheduled to undergo elective surgical procedures or heathy control. 150 participants will be recruited in total.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with full stomach | one day
  The main objective is to compare the frequency of a "full stomach" in the diabetic population compared to a healthy control population 2h after clear liquid or 6h after light meal.

SECONDARY OUTCOMES:
the mean gastric emptying time of clear liquid and light meal | one day
  To assess the mean gastric emptying time of clear liquid and light meal in the diabetic population

OTHER OUTCOMES:
Correlation of diabetes mellitus complications with delayed stomach empty | one day
  To assess whether there is significant correlation between diabetes mellitus related eye disease, cardiovascular cardiovascular autonomic neuropathy, peripheral neuropathy (MNSI) with delayed stomach empty

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided